CLINICAL TRIAL: NCT02209454
Title: Comparative Study of the Bioavailability of Dexketoprofen Trometamol Following Single Doses of 25mg Enantyum® Oral Solution vs. Keral® Tablets in Healthy Subjects
Brief Title: Comparative Bioavailability of Dexketoprofen Trometamol Oral Solution vs Tablet Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Menarini Group (Industry)
Collaborators: Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: RD 303/25652(DKP-BE-SOL); 2014-000371-10 (EudraCT Number)
Record Dates: First submitted 2014-08-04; First posted 2014-08-06 (Estimated); Results first posted 2015-07-09 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-05

CONDITIONS: Acute Pain
Keywords: Dexketoprofen; Bioavailability; Comparative; Pharmacokinetic
MeSH Terms: conditions — Acute Pain | interventions — dexketoprofen trometamol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enantyum® oral solution (Other): 25mg DKP.TRIS oral solution
  Interventions: Drug: Enantyum® oral solution
- Keral® tablet (Other): 25mg DKP.TRIS tablet
  Interventions: Drug: Keral® tablet

INTERVENTIONS:
Drug: Enantyum® oral solution — One dose of 25 mg DKP oral solution
  Arms: Enantyum® oral solution
Drug: Keral® tablet — One dose of 25 mg DKP tablet
  Arms: Keral® tablet

SUMMARY:
The purpose of this study is to compare the bioavailability of 25 mg DKP.TRIS given as an Enantyum® oral solution (Test formulation) and Keral® tablet (Reference formulation). In addition, this study intends to evaluate the safety and tolerability of Test and Reference formulations.

DETAILED DESCRIPTION:
The study was conducted in 1 site and included 26 successfully screened and randomized healthy subjects(12 female and 14 male).

The study consisted of:

* Screening Visit (performed within 3 weeks prior to 1st PK study session), for the evaluation of study eligibility.
* Two pharmacokinetic (PK) study sessions, separated by a minimum of a 7 day washout period, including the administration of one out of 2 study treatments at each study session (namely 25mg DKP.TRIS given as Enantyum® oral solution or Keral® tablet) according to the sequence as per randomisation list, and blood sampling for PK assessment on plasma at pre-defined time up to 24 hours post-dose.
* End of Study Visit (7-10 days after last treatment administration).

ELIGIBILITY:
Inclusion Criteria:

- Healthy male and female subjects between 18 to 50 years old, with a Body Mass Index (BMI) between 18 Kg/m2 and 28 Kg/m2-

Exclusion Criteria:

* History of previous allergy idiosyncrasy / sensitivity to DKP.TRIS or other NSAIDs (aspirin, ibuprofen etc).
* Any condition which might interfere with the absorption, distribution, metabolism or excretion of the drugs.
* Surgery within previous 6 months, or blood loss > 400 mL within previous 3 months.
* Subject with positive human immunodeficiency virus (HIV), hepatitis B surface antigen (Hep B) and hepatitis C virus antibody (Hep C) results.
* History of clinically significant alcohol, medicine or drug abuse.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Girish Sharma, MBBS, Principal Investigator — Simbec Research
Locations (1):
- Simbec Research Limited, Merthyr Tydfil, UK, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Reference IMP First, Then Test IMP: 25mg DKP.TRIS tablet one single administration in first period and 25mg DKP.TRIS oral solution one single administration in second period (after washout period).
- Test IMP First, Then Reference IMP: 25mg DKP.TRIS oral solution one single administration in first period and 25mg DKP.TRIS tablet one single administration in second period (after washout period).
Period: First Period
Arm/Group | Reference IMP First, Then Test IMP | Test IMP First, Then Reference IMP
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0
Period: Washout Period a Minimum of a 7 Day
Arm/Group | Reference IMP First, Then Test IMP | Test IMP First, Then Reference IMP
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0
Period: Second Period
Arm/Group | Reference IMP First, Then Test IMP | Test IMP First, Then Reference IMP
Started | 13 | 13
Completed | 12 | 13
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Twenty-six (26) subjects were randomized (14 male and 12 female) for 24 to complete the study. A total of 25 subjects (13 male and 12 female) completed the study. NOTE: Treatments were administered in a crossover manner, with the same population but one healthy subjects being exposed to the Reference and Test IMP.
Groups:
- Entire Study Population: Includes groups randomized to receive 25mg DKP.TRIS tablet first and 25mg DKP.TRIS oral solution first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.9 (6.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 14
Region of Enrollment [Number; unit: participants]
  United Kingdom | 26

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: The absence of any difference in the rate and extent of absorption will be demonstrated if the 90% CI for the geometric mean ratio between Test and Reference formulations is within the range 80.00% - 133.00% for Cmax.
Time Frame: Up to 24h post-dose (pre-dose, T+5', T+10', T+15', T+20', T+30', T+40', T+50', T+1h, T+1.25h, T+1.5h, T+2h, T+3h, T+3.5h, T+4h, T+5h, T+6h, T+8h, T+12h and T+24h post-dose).
Population: Analyses of the primary PK variables were conducted on all randomised subjects who received at least one dose of DKP.TRIS (PK population) and on all subjects in the PK population who did not experience major protocol violations (PP population).
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Enantyum® Oral Solution | Keral® Tablet
Number analyzed (Participants) | 25 | 26
ng/mL | 3290.70 [2996.00 to 3614.40] | 2785.90 [2493.20 to 3113.00]

2. Secondary Outcome: AUC(0-∞)
Description: AUC(0-∞) will be analysed similarly to AUC(0-t) and Cmax. Time to achieve maximum plasma concentration (tmax) and t1/2 will be summarized descriptively.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Enantyum® Oral Solution | Keral® Tablet
Number analyzed (Participants) | 25 | 26
h*ng/mL | 3473.00 [3087.70 to 3906.40] | 3485.60 [3135.30 to 3875.00]

3. Primary Outcome: AUC(0-t)
Description: The absence of any difference in the rate and extent of absorption will be demonstrated if the 90% CI for the geometric mean ratio between Test and Reference formulations is within the range 80.00% - 125.00% for AUC(0-t).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Enantyum® Oral Solution | Keral® Tablet
Number analyzed (Participants) | 25 | 26
h*ng/mL | 3362.20 [2986.20 to 3785.60] | 3372.00 [3027.30 to 3755.90]

4. Secondary Outcome: Tmax
Description: AUC(0-∞) will be analysed similarly to AUC(0-t) and Cmax. Time to achieve maximum plasma concentration (tmax).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Enantyum® Oral Solution | Keral® Tablet
Number analyzed (Participants) | 25 | 26
h | 0.25 [0.17 to 0.67] | 0.50 [0.25 to 1.25]

5. Secondary Outcome: t1/2
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: h
Arm/Group | Enantyum® Oral Solution | Keral® Tablet
Number analyzed (Participants) | 25 | 26
h | 1.34 [1.23 to 1.45] | 1.30 [1.20 to 1.41]

ADVERSE EVENTS:
Time Frame: from Screening Visit to End of Study Visit
Description: Analyzed for the safety population (All subject receiving at least one administration of study treatment)
Arm/Group | Enantyum® Oral Solution | Keral® Tablet
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 4/25 | 7/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enantyum® Oral Solution (N=25) | Keral® Tablet (N=26)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (2)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Serum ferritin decreases (Investigations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No